CLINICAL TRIAL: NCT03644121
Title: Adherence to Continuous Positive Airway Pressure in Patients With Obstructive Sleep Apnoea Syndrome. Ten Year Follow up
Brief Title: Adherence to CPAP in Patients With OSA. Ten Year Follow up
Status: Completed | Type: Observational
Sponsor: Maugeri Foundation (Other)
Responsible Party: Principal Investigator, elisabetta zampogna, principal investigator, Maugeri Foundation
Other Study IDs: 2215CE
Record Dates: First submitted 2018-07-10; First posted 2018-08-23 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: OSA; Adherence, Patient; CPAP
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The management of OSA is aimed to improve symptoms and mitigate reduce other health consequences. Continuous Positive Airway Pressure (CPAP) is the recognized treatment for OSA, able to reverse the pathophysiology of OSA and improving sleep continuity, resulting in improvements in daytime sleepiness and quality of life (QoL). However, low adherence to this treatment reduces the potential to achieve these benefits. The aim of this real life retrospective observational study was to assess the adherence to CPAP at 12 month and 10 years. The investigators evaluated also predicitve factors of adherence.

DETAILED DESCRIPTION:
Methods The protocol was approved (2215 CE, June, 19, 2018) by the Ethical Committee of the Istituti Clinici Scientifici (ICS) Maugeri, Pavia, Italy. All patients at admission to the Scientific Institute of Tradate gave the informed consent to the scientific use of their data.

Study Participants This study was conducted on a database of patients' discharge records, available between August, 2006 and December, 2009.

Adaptation to CPAP: titration of CPAP was performed either by full-night manual titration according to the AASM Guidelines or by automatic titration with Auto-Set systems. Further 4 day-time hours of adaptation were performed along two days. Patients underwent also four face to face sessions with the respiratory therapist, for feed-back of adaptation, optimal comprehension of procedure of CPAP management. The presence of a caregiver (if any) was strongly suggested.

Statistical Analysis An ad hoc electronic form was created to collect all study variables. Qualitative variables were described with absolute and relative (percentages) frequencies, whereas quantitative variables were summarized with means (standard deviations) or medians (interquartile ranges) based on their normal distribution, respectively.

In-between comparison for qualitative and quantitative variables was performed with the chi-squared or Fisher exact test when appropriate, and Student t or Mann-Whitney test in case of parametric or non-parametric distribution, respectively. Comparison of the temporal variation of continuous variables for the same group was assessed with Anova or Friedman's test, depending on their normal distribution.

Uni- and multi-variable logistic regression analysis was performed to assess which covariates could be associated with the adherence to CPAP.

A two-tailed p-value <0.05 was considered significant. All statistical analyses were carried out using the statistical software STATA version 15 (StatsCorp, Texas).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of OSA
* admitted for adaptation to CPAP

Exclusion Criteria:

* other sleep related diseases
* concomitant lung or thoracic diseases (including chronic respiratory failure requiring long term oxygen therapy)
* major comorbidities (e.g. psychiatric conditions, cancer, end-stage renal failure)
* familiar conditions preventing long-term home CPAP
* patients already treated with CPAP

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diagnosis of OSA. According to the International Classification of Sleep Disorders, OSA was defined as the presence of 5 or more obstructive respiratory events (apnea, hypopnea or respiratory effort-related arousal) per hour of sleep plus daytime or nighttime symptoms of OSA, alternatively as the presence of 15 or more obstructive respiratory events per hour of sleep
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2006-08-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-06 (Actual)

PRIMARY OUTCOMES:
CPAP use | Every 12 month for 10 years.Scale from 0 to 8 hours/night. Values >4,5 hours/night are considered to be a better outcome
  number of Night-time hours of use (device counter)

SECONDARY OUTCOMES:
Body weight | once a year for 10 years
  Kg
Reported patients' day-time sleepiness | once a year for 10 years
  Epworth Sleepness Scale (ESS).The questionnaire asks the subject to rate his/her probability of falling asleep on a scale of increasing probability from 0 to 3 for eight different situations that most people engage in during their daily lives. The scores for the eight questions are added together to obtain a single number. A number in the 0-9 range is considered to be normal while a number in the 10-24 range indicates that expert medical advice should be sought

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Spanevello, Prof MD, Study Director — Maugeri Foundation, Insubria University
Locations (1):
- Maugeri Foundation, Tradate, VA, Italy

IPD SHARING:
Plan to Share IPD: Yes
Publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 4 month
Access Criteria: free